CLINICAL TRIAL: NCT06686342
Title: Consistency Evaluation of Drug Efficacy Between Clinical Systemic Treatment and Drug Sensitive Test Based on Patient-derived Organoid in Patients With Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma: A Prospective, Multicenter, Observational Study
Brief Title: PDO Based Drug Sensitive Test in R/M HNSCC
Status: Recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Collaborators: Shanghai Cancer Hospital, China (Other); Eye & ENT Hospital of Fudan University (Other); Dongfang Hospital Affiliated to Tongji University (Other); Shandong Cancer Hospital and Institute (Other); Qilu Hospital of Shandong University (Other); Shandong Provincial Hospital (Other Government); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Tongji Hospital (Other); Hospital of Stomatology, Wuhan University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); First Affiliated Hospital of Zhejiang University (Other); Sir Run Run Shaw Hospital (Other); Zhejiang Cancer Hospital (Other); Shanghai Zhongshan Hospital (Other); Shanghai Huangpu District Central Hospital (Unknown)
Responsible Party: Principal Investigator, Lai-ping Zhong, Professor, Huashan Hospital
Other Study IDs: DST-PDO-HNSCC
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Patient Derived Organoid; Drug Sensitive Test in Vitro
Keywords: Recurrent/metastatic head and neck squamous cell carcinoma; Patient-derived organoid; Drug sensitive test in vitro
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational cohort: The observational group of patients with R/M HNSCC would receive drug treatment according to the clinical guideline or doctor's experience. No intervention would be provided based on the drug sensitive test from patient-derived organoid.
  Interventions: Other: No intervention; Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No intervention — The patients with R/M HNSCC would receive drug treatment according to the clinical guideline or doctor's experience, at the same time, tumor biopsy samples would be collected to establish PDO for drug sensitive test. But no intervention would be used based on the PDO drug sensitive test.
Other: No Intervention: Observational Cohort — The patients with R/M HNSCC would receive drug treatment according to the clinical guideline or doctor's experience, at the same time, tumor biopsy samples would be collected to establish PDO for drug sensitive test. But no intervention would be used based on the PDO drug sensitive test.

SUMMARY:
To evaluate the consistency of drug efficacy between the clinical systemic treatment and drug sensitive test based on patient-derived organoid in R/M HNSCC patients, using a prospective and multicenter observational study to increase the generalizability and reliability of research conclusion.

DETAILED DESCRIPTION:
Head and neck squamous cell carcinoma (HNSCC) is one of the most common cancers threatening human health, recurrent and metastatic HNSCC (R/M HNSCC) is the most difficult to treat, and the prognosis is very poor. Drug treatment is the mostly choice; however, individualized treatment needs to determine the specific treatment plan according to the characteristics of the patient and the tumor. In addition to NGS sequencing, high-throughput models for in vitro drug sensitive tests are an effective means to improve clinical efficacy.

Organoids are in vitro cultured micro-organs with 3D structures, capable of spontaneous self-renewal, self-organization, and differentiation to form complex structures similar to real tissues, partially simulating the physiological functions of the source tissue or organ. Compared with other in vitro and in vivo models such as cell lines and patient-derived xenograft models, organoid models have unique advantages: they can more vividly retain the phenotypic, genetic, and functional characteristics of the original tissue, and have a short modeling cycle, high cost-performance ratio, and can achieve high throughput drug sensitive test. In 2018, a study showed that ex vivo drug sensitivity testing based on gastrointestinal tumor organoids has a very high predictive value for clinical efficacy, with a sensitivity of 100%, specificity of 93%, and positive and negative predictive values of 88% and 100%, respectively. In addition, cancer organoids have been developed from many other cancer types and its feasibility in guiding precision medicine is investigated. The aim of present study is to evaluate the consistency of drug efficacy between the clinical systemic treatment and drug sensitive test based on patient-derived organoid in R/M HNSCC patients. A prospective and multicenter observational study is planned to increase the generalizability and reliability of research conclusion.

The patients with R/M HNSCC would receive drug treatment according to the clinical guideline or doctor's experience, at the same time, tumor biopsy samples would be collected to establish PDO for drug sensitive test. Fifteen different drug regimens sensitive test would be performed, including the actual drug regimens that the patients clinically receive, and the corresponding ex vivo tumor inhibition rate would be recorded. After the patients received the clinical treatment, they would be followed up to collect the objective response rate (ORR), disease control rate (DCR), progression-free survival time (PFS), and overall survival time (OS). Finally, the consistency of drug efficacy would be evaluated between clinical systemic treatment and drug sensitive test based on patient-derived organoid.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed R/M HNSCC patients
* Tumor tissues available for organoid culture
* ECOG score: 0-2 points
* Life expectancy > 3 months
* Normal major organ function, tolerable to chemotherapy, targeted therapy, immunotherapy: a. Hematology examination criteria must meet: WBC≥4.0×109/L, ANC≥1.5×109/L, PLT≥80×109/L, Hb≥90 g/L (no blood transfusion or blood products within 14 days, no use of G-CSF or other hematopoietic growth factors); b. Biochemical examination must meet the following criteria: serum albumin≥3.0 g/dL (30 g/L), TBIL≤1.5×ULN, ALT, AST≤2.5×ULN, BUN and CRE≤1.5×ULN or endogenous creatinine clearance≥60 ml/min (Cockcroft-Gault formula); c. Good coagulation function: defined as International Normalized Ratio (INR) or Prothrombin Time (PT)≤1.5 times ULN; if the study participant is on anticoagulant therapy, as long as PT is within the intended range of the anticoagulant medication
* Able to understand the content of informed consent form, sign the informed consent form, and willing to cooperate with the follow-up

Exclusion Criteria:

* Metastatic tumors in the head and neck region, or non-HNSCC such as sarcoma, adenocarcinoma, nasopharyngeal carcinoma, etc.
* Known allergy to the study drugs or their active ingredients or any excipients; or had a severe allergic reaction to other monoclonal antibodies
* Pregnant or breastfeeding female patients; or women of childbearing age with positive pregnancy test results (serum or urine) within 7 days before enrollment, or negative results but refusing to use effective contraception during the study period and 2 months after the last administration of study medication; or male patients with partners of childbearing age, refusing to use effective contraception during the study period and 2 months after the last administration of study medication
* Severe liver diseases (such as cirrhosis), kidney diseases, respiratory system diseases, hematopoietic system diseases, or endocrine system diseases, uncontrolled diseases
* Infected with HIV, active hepatitis B (HBV-DNA≥104 copies/ml) or hepatitis C (hepatitis C antibody positive, and HCR-RNA above the lower limit of detection of the analytical method), uncontrolled diseases
* Within 6 months before enrollment, the following conditions occurred: myocardial infarction, severe/unstable angina, NYHA class 2 or above heart failure, clinically significant supraventricular or ventricular arrhythmias, and symptomatic congestive heart failure, uncontrolled diseases
* Patients with mental illness or known history of psychiatric drug abuse or drug addiction
* Unable to give consent, unable to obtain the required amount of tumor tissue for the study
* Other serious physical or mental diseases or laboratory test abnormalities that may increase the risk of participating in the study or interfere with the study results; or any other situation that the researchers deem unsuitable for participation in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is an observational study, according to previous literature reports combined with the actual clinical situation of institution/collaborating institutions, a total of 100 participants are planned to be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2026-11-11 (Estimated); Study Completion 2028-11-11 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 2 years
  The proportion of patients whose tumor size is reduced to a pre-specified value and maintained for a minimum required duration, which is the sum of the proportions of Complete Response (CR) and Partial Response (PR).
Disease Control Rate | 2 years
  The proportion of patients whose tumor size is reduced or stable and maintained for a minimum required duration, which is the sum of the proportions of Complete Response (CR), Partial Response (PR), and Stable Disease (SD).

SECONDARY OUTCOMES:
The success rate of establishment and drug sensite test on PDO | 2 years
  Number of successful organoid construction and completion of drug sensitive test/Total number of participants ×100%.
Tumor Growth Inhibition of PDO | 2 weeks
  (1-T/C) × 100%, where T is the survival rate of PDO drug treatment group, and C is the survival rate of PDO control group.
Overall Survival | 2 years
  The time from enrollment of participants to death (for any reason).
Progression-Free Survival | 2 years
  The time from enrollment of participants to occurrence of tumor progression (in any aspect) or death (for any reason).

CONTACTS AND LOCATIONS:
Overall Officials: Lai-ping Zhong, MD, PhD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
After the completion of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2 years after completion of the study, for 6 months.
Access Criteria: Access to IPD data can be obtained upon scientifically sound request from the study PI, who will contact the Clinical Research Unit, Huashan Hospital, Fudan University. Access will be released after the approval from the Clinical Research Unit.

REFERENCES:
- [Background] Pasch CA, Favreau PF, Yueh AE, Babiarz CP, Gillette AA, Sharick JT, Karim MR, Nickel KP, DeZeeuw AK, Sprackling CM, Emmerich PB, DeStefanis RA, Pitera RT, Payne SN, Korkos DP, Clipson L, Walsh CM, Miller D, Carchman EH, Burkard ME, Lemmon KK, Matkowskyj KA, Newton MA, Ong IM, Bassetti MF, Kimple RJ, Skala MC, Deming DA. Patient-Derived Cancer Organoid Cultures to Predict Sensitivity to Chemotherapy and Radiation. Clin Cancer Res. 2019 Sep 1;25(17):5376-5387. doi: 10.1158/1078-0432.CCR-18-3590. Epub 2019 Jun 7. PMID 31175091
- [Background] Vlachogiannis G, Hedayat S, Vatsiou A, Jamin Y, Fernandez-Mateos J, Khan K, Lampis A, Eason K, Huntingford I, Burke R, Rata M, Koh DM, Tunariu N, Collins D, Hulkki-Wilson S, Ragulan C, Spiteri I, Moorcraft SY, Chau I, Rao S, Watkins D, Fotiadis N, Bali M, Darvish-Damavandi M, Lote H, Eltahir Z, Smyth EC, Begum R, Clarke PA, Hahne JC, Dowsett M, de Bono J, Workman P, Sadanandam A, Fassan M, Sansom OJ, Eccles S, Starling N, Braconi C, Sottoriva A, Robinson SP, Cunningham D, Valeri N. Patient-derived organoids model treatment response of metastatic gastrointestinal cancers. Science. 2018 Feb 23;359(6378):920-926. doi: 10.1126/science.aao2774. PMID 29472484